CLINICAL TRIAL: NCT06515587
Title: To Evaluate a Prospective, Multicenter, Exploratory Clinical Study of Lewis Antigen Assay Combined With CA19-9 Assay to Assess Prognosis in Patients With Pancreatic Cancer
Brief Title: Clinical Study of Lewis Antigen Assay Combined With CA19-9 Assay to Assess Prognosis in Patients With Pancreatic Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiang Long, Head of pancreatic surgery, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Lewis-IIT-202401
Record Dates: First submitted 2024-06-25; First posted 2024-07-23 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: PDAC

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): All enrolled subjects will accurately complete one Lewis genotype test and at least one CA19-9 test
  Interventions: Diagnostic Test: Lewis genotype detection reagent

INTERVENTIONS:
Diagnostic Test: Lewis genotype detection reagent — By evaluating the results of the Lewis gene test combined with the CA19-9 test, different subtypes of pancreatic cancer patients were differentiated to evaluate the prognosis

SUMMARY:
CA19-9 is an acidic glycoside containing sialic acid, called ganglioside. Lewis blood group antigen is the precursor for the synthesis of CA19-9, which is formed by the combined action of sialic acid transferase and fucosyltransferase (FUT3). The ability to produce soluble blood group substances is determined by the alpha (1,2) fucosyltransferase gene (FUT2), which can be divided into secretory Se, weakly secretory Sew, and non secretory SE. The Lewis antigen positive (Lewis+) population has normal CA19-9 secretion function, while the Lewis antigen negative (Lewis -) population (about 7%) usually shows no or low secretion of CA19-9. Therefore, when CA19-9 is used as a biomarker, the combined detection of Lewis antigen status is a marker to judge the prognosis of pancreatic cancer, which can divide pancreatic cancer patients into high/medium/low malignant phenotypes.

DETAILED DESCRIPTION:
1. This study adopts a prospective, multicenter design, and classifies pancreatic cancer patients and predicts their prognosis through Lewis antigen detection and CA19-9 detection.
2. Observe the survival time of pancreatic cancer subjects to observe the consistency between Lewis typing and prognosis, and evaluate the sensitivity of Lewis antigen detection.
3. Evaluate the specificity of Lewis antigen detection by observing the distribution of Lewis subtypes in non pancreatic cancer subjects.
4. Explore the prognostic distribution of age, different Lewis subtypes, and overall survival cycle for Lewis antigen detection.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily enrolled, regardless of gender, aged ≥ 18 and ≤ 75 years old, and the patient can understand and is willing to sign an informed consent form;
2. ECOG 0-2
3. Pathologically confirmed as pancreatic ductal adenocarcinoma; Or confirmed by pathology and clinical examination as pancreatic ductal adenocarcinoma.
4. Willing to accept routine CA19-9 testing, Lewis antigen sample collection and testing (2-3ml), and follow-up Non pancreatic cancer subjects enrolled in this study must meet all the following criteria

1. Voluntary enrollment, regardless of gender, age ≥ 18 years, ≤ 75 years old, and the patient can understand and is willing to sign an informed consent form 2. Willing to accept Lewis antigen sample collection and testing (2-3ml)

Exclusion Criteria:

1. Suffering from the second or double primary malignant tumor besides pancreatic cancer at the same time
2. Patients with pancreatic cancer who cannot trace the specific anti-cancer treatment plan
3. HIV positive
4. Other situations that researchers believe need to be excluded

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
To explore the prognosis of pancreatic cancer with the combination of the Lewis antigen test and the CA19-9 test | Up to 12 months after the treatment
  The phenotypes of pancreatic cancer patients were classified by Lewis antigen test combined with CA19-9 test.Monitoring patients' disease expression and assisting clinical selection of targeted treatment plan.The consistency between Lewis classification and prognosis was assessed by looking at the survival of pancreatic cancer subjects following clinical treatment regimens.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China